CLINICAL TRIAL: NCT06875921
Title: Home-Based, Video-Supported McKenzie vs. Pilates Exercise Programs for Individuals With Chronic Low Back Pain
Brief Title: McKenzie vs Pilates Exercises in People With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Hellenic University (Other)
Responsible Party: Principal Investigator, Dimitrios Lytras, Assistant Professor, International Hellenic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC-7 2025
Record Dates: First submitted 2025-03-09; First posted 2025-03-13 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-03

CONDITIONS: Chronic Low Back Pain
Keywords: Chronic low back pain; Pilates; McKenzie; Physiotherapy; Home-based exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: A masked assessor will conduct the measurements
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- McKenzie Exercises (Experimental): Participants allocated to this group will perform exercises based on the McKenzie Method at home, once a day for three weeks.
  Interventions: Other: McKenzie Exercise Group
- Pilates Exercises (Experimental): Participants allocated to this group will perform exercises based on the Pilates Method at home, twice a week for three weeks.
  Interventions: Other: Pilates Exercise Group

INTERVENTIONS:
Other: McKenzie Exercise Group — The intervention will last 7 minutes and will consist of the following exercises:
  * Four Extension Exercises: Lying Face Down, Lying Face Down in Extension, Repeated Lumbar Extension in Lying, Repeated Lumbar Extension in Standing.
  * Two Flexion Exercises: Repeated Lumbar Flexion in Lying, Repeated Lumbar Flexion in Sitting.
  Arms: McKenzie Exercises
Other: Pilates Exercise Group — The intervention will last 20 minutes and will include Pilates exercises focused on mobility and strengthening.
  Arms: Pilates Exercises

SUMMARY:
Brief Summary: Chronic low back pain (CLBP) is a persistent condition lasting more than 12 weeks, often leading to pain, disability, and reduced quality of life. This clinical study aims to compare the effectiveness of McKenzie and Pilates exercise programs in managing CLBP symptoms. A total of 32 participants will be randomly assigned to two equal groups: one performing McKenzie exercises and the other engaging in Pilates routines. The intervention will span three weeks. Outcomes will be assessed using the Visual Analogue Scale (VAS) for pain intensity, the Roland-Morris Disability Questionnaire (RMDQ) for functional impairment, a pressure algometer for pain sensitivity (PPT), and the Fingertip-to-Floor test (FTF) for range of motion (ROM). A two-way repeated-measures ANOVA will be used for statistical analysis, with significance set at p < .05.

DETAILED DESCRIPTION:
Background Chronic low back pain (CLBP) is characterized by persistent pain in the lumbar region lasting for more than 12 weeks, often leading to functional limitations and a decline in quality of life. Exercise-based interventions, such as the McKenzie method and Pilates, are widely implemented in managing CLBP symptoms, but direct comparisons of their effectiveness remain limited.

Aim This study aims to evaluate and compare the effects of the McKenzie method and Pilates exercises on pain relief, functional disability, and range of motion in individuals with CLBP. The objective is to determine whether one approach is more beneficial than the other in alleviating symptoms and enhancing physical function.

Method Thirty-two participants diagnosed with CLBP will be randomly assigned into two equal groups. One group will follow a McKenzie-based exercise program, while the other will engage in a Pilates regimen. Both interventions will last three weeks. Pain intensity will be assessed using the Visual Analogue Scale (VAS), functional disability will be measured with the Roland-Morris Disability Questionnaire (RMDQ), pain sensitivity will be evaluated through the pressure pain threshold (PPT) using an algometer, and range of motion will be determined by the Fingertip-to-Floor (FTF) test. Measurements will be taken before and after the intervention. Statistical analysis will be conducted using a two-way repeated-measures ANOVA to examine within- and between-group differences, with the significance level set at p < .05.

Expected Results This study aims to compare the effectiveness of McKenzie and Pilates exercises in managing CLBP symptoms. Both methods are expected to provide significant improvements in pain reduction, disability, and pain sensitivity. However, since Pilates exercises emphasize flexibility, it is anticipated that they will result in a greater improvement in range of motion compared to the McKenzie method. Consequently, while similar outcomes are expected in most measured parameters, a superior increase in ROM is anticipated in the Pilates group.

ELIGIBILITY:
Inclusion Criteria:

* Duration of symptoms 12 weeks
* Age range between 18 and 60 years
* Pain score ≥ 2cm in VAS scale
* Written consent to participate in the study

Exclusion Criteria:

* Neuropathic pain extending along the lower limb due to nerve root compression
* Previous spine surgery
* History of spine trauma or fracture
* Implanted pacemakers
* Pregnancy
* Cancer
* Systemic musculoskeletal diseases, diagnosed neurodegenerative diseases (e.g., Parkinson's), epilepsy, and history of psychiatric disorders

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-04-20 (Actual); Study Completion 2025-04-20 (Actual)

PRIMARY OUTCOMES:
Changes in Low Back Pain (LBP) Intensity Using the Visual Analog Scale (VAS) | Pre-treatment, Post-treatment (Week 3)
  The VAS is a 10 cm pain scale with no numerical markings. The left end represents "No pain," while the right end corresponds to "Worst possible pain." A higher score indicates greater pain intensity. Participants will complete the scale twice-before and after the intervention-marking the level of pain experienced over the past 24 hours. Pain intensity will be quantified by measuring the distance from the zero point ("No pain") to the indicated score
Changes in Pressure Pain Threshold (PPT) Using Pressure Algometry | Pre-treatment, Post-treatment (Week 3)
  Pressure pain threshold (PPT) refers to the minimum amount of pressure required to elicit pain. A digital algometer will be used to measure PPT bilaterally at the L4-L5 intervertebral space. The device's metal rod will be placed perpendicularly on the site, and pressure will be gradually increased at a rate of 1 kg/s until the participant reports pain. PPT will be recorded in N/cm².
Changes in Functional Capacity Using the Greek Version of the Roland-Morris Disability Questionnaire (RMDQ) | Pre-treatment, Post-treatment (Week 3)
  Functional capacity will be assessed using the validated Greek version of the Roland-Morris Disability Questionnaire (RMDQ), which consists of 24 items addressing daily activities impacted by low back pain. Each selected statement adds one point to the total score, with higher values indicating greater disability.
4. Changes in Lumbar Spine Flexion Range of Motion Using the Fingertip-to-Floor (FTF) Test | Pre-treatment, Post-treatment (Week 3)
  Spinal mobility will be evaluated using the Fingertip-to-Floor Test, a widely used clinical tool for assessing trunk flexion. Participants will be asked to bend forward and reach toward the ground while keeping their knees and hips extended. The examiner will measure the vertical distance between the participant's fingertips and the floor using a tape measure.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physiotherapy, Faculty of Health Sciences International Hellenic University, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No